CLINICAL TRIAL: NCT02458963
Title: In Vitro Fertilization Versus Gonadotropin Therapy in Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome
Brief Title: IVF Versus Gonadotropin Therapy in Women With CC Resistant PCOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG3
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infertility; Polycystic Ovarian Syndrome
Keywords: PCOS; Clomiphene citrate resistant; Gonadotropin; IVF
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Sperm Injections, Intracytoplasmic; Gonadotropins; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVF group (Active Comparator): Women will undergo one full IVF cycle
  Interventions: Procedure: IVF
- Gonadotropin group (Active Comparator): Women will be subjected to ovarian stimulation for 6 months with the gonadotropin low-dose step-down protocol.
  Interventions: Drug: Gonadotropin

INTERVENTIONS:
Procedure: IVF — Women will undergo one IVF cycle
  Other Names: Intracytoplasmic sperm injection (ICSI)
  Arms: IVF group
Drug: Gonadotropin — Women will be subjected to ovarian stimulation for 6 months with the gonadotropin low-dose step-down protocol
  Other Names: Human Menopausal Gonadotropin (HMG)
  Arms: Gonadotropin group

SUMMARY:
The purpose of this study is to compare the efficacy of in vitro fertilization (IVF) versus gonadotropin therapy in infertile women having clomiphene citrate (CC) resistant polycystic ovarian syndrome (PCOS).

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; IVF group and gonadotropin group. Women in the IVF group will undergo one full IVF cycle. Women in the gonadotropin group will be subjected to ovarian stimulation for 6 months with the gonadotropin low-dose step-down protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with PCOS as defined by the Rotterdam criteria.
* CC resistance (defined as failure of ovulation after receiving 150 mg/day of CC for 5 consecutive days per cycle, for at least 3 consecutive cycles).

Exclusion Criteria:

* Age < 20 or > 35 years.
* Presence of any infertility factor other than anovulatory PCOS.
* Previous history of ovarian surgery or surgical removal of one ovary.
* Previous exposure to cytotoxic drugs or pelvic irradiation.
* Oral hypoglycemic or hormonal therapy either currently or in the preceding 3 months.
* Metabolic or hormonal abnormalities.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 9 months
  Number of live births divided by the number of women

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6-8 weeks gestational age
  Number of clinical pregnancies divided by the number of women
Multifetal pregnancy rate | 12 weeks gestational age
  Number of multifetal pregnancies divided by the number of clinical pregnancies
Miscarriage rate | 12 weeks gestational age
  Number of first trimester miscarriages (before 12 weeks gestational age) divided by the number of clinical pregnancies
Incidence of early ovarian hyperstimulation syndrome (OHSS) | Within 9 days of final triggering of oocyte maturation
  Incidence of OHSS within 9 days of final triggering of oocyte maturation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, Dr, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University
Locations (2):
- Egypt (2):
  - Fertility Care Unit (FCU) in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private fertility care centers, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Undecided